CLINICAL TRIAL: NCT05954845
Title: The Enteric Nervous System in Spinal Cord Injury : étude du système Nerveux entérique et de la barrière épithéliale Intestinale Via la réalisation de Biopsies Coliques Chez Les Patients Porteurs de lésion médullaire
Brief Title: The Enteric Nervous System in Spinal Cord Injury: Study of the Enteric Nervous System and the Intestinal Epithelial Barrier Via Colonic Biopsies in Spinal Cord Injury Patients
Acronym: TENS-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC23_0075
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury, Neurogastroenterology, Pathophysiology, Enteric nervous system, Intestinal epithelial barrier
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: participants will have colonic biopsies taken following a colonoscopy/rectosigmoidoscopy previously indicated. Biopsies will be obtained from the right and left colon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with spinal cord injury (Experimental)
  Interventions: Other: biopsies
- Control (Other): Patients with no spinal cord injury
  Interventions: Other: biopsies

INTERVENTIONS:
Other: biopsies — Biopsies will be obtained from the right and left colon (5 biopsies per colic region)

SUMMARY:
The goal of this clinical trial is to learn more about the enteric nervous system (ENS) and the intestinal epithelial barrier (IEB) in patients with spinal cord injury (SCI). The main questions it aims to answer are :

* to characterize the functional (permeability, serotonin production, enteric neuronal phenotype, etc.), proteomic (junction molecules) and transcriptomic (inflammation genes, neuromediator expression, etc.) remodeling of the colonic mucosa and ENS in SCI patients, in comparison with control data.
* to correlate intestinal permeability (and all remodeling parameters) with the type of neurological impairment i.e. the neurological level of the lesion, quantification of neurological impairment (motor and sensory scores) and the completeness and incompleteness of a lesion.
* to identify a link with disease severity markers
* to identify therapeutic targets that could subsequently be tested in the animal model before being proposed in clinical trials.

Participants will have colonic biopsies taken following a colonoscopy/rectosigmoidoscopy previously indicated for spinal cord injured patients. Biopsies will be obtained from the right and left colon.

DETAILED DESCRIPTION:
Injury to the spinal cord, whether traumatic or not, leads to numerous organ deficiencies, particularly vegetative deficiencies. Digestive and anorectal dysfunctions are among these, and are the main deficiencies that spinal cord injury patients would like to see disappear, even before motor recovery or walking, for example. However, the treatments available are essentially empirical (dietary hygiene rules, use of laxatives, digital exoneration maneuvers) and only partially effective.

Pathophysiological knowledge of digestive dysfunction in the medullo-injured is mainly focused on dysfunctions of extrinsic vegetative innervation. In contrast, there are few studies concerning the dysfunction of intrinsic digestive innervation in this pathology, i.e. the enteric nervous system (ENS), and the intestinal epithelial barrier (IEB), which are central players involved in the digestive disorders observed during the course of numerous digestive or extra-digestive pathologies, such as Parkinson's Disease (PD) in particular.

To date, the nature of ENS/EIB remodeling has not been correlated with clinical data, in order to potentially link it to a clinical phenotype of these patients, and to determine their capacity to become predictive biomarkers of disease progression, severity and/or response to treatment. By combining functional exploration of the intestinal barrier, protein and transcriptomic analysis of biopsies, the aim is to 1) characterize functional (permeability, serotonin production), proteomic and transcriptomic remodeling of the mucosa in SCI patients compared with control groups, 2) make the link with patients' clinical data, 3) identify markers of disease severity (lesion level, severity of intestinal dysfunction) and 4) identify therapeutic targets that could be tested in the animal model before being proposed in clinical trials.

ELIGIBILITY:
Inclusion Criteria for patient with spinal cord injury:

Patient with signed consent Patient over 18 and under 80 years of age Patient with acquired traumatic or non-traumatic spinal cord injury Patient with an indication for colonoscopy or rectosigmoidoscopy at the Nantes University Hospital Gastroenterology Department Eligible for French social security Patient enrolled in the COSCINUS cohort

Inclusion criteria for control group:

Subject with signed consent Subject over 18 and under 80 years of age Subject free of any neurological pathology, with an indication for screening or preventive colonoscopy in the context of a personal or family history of polyps, or familial colon cancer, in the gastroenterology department of the Nantes University Hospital.

Exclusion Criteria for patients with spinal cord injury:

Patients in emergency situations, deprived of liberty, or not covered by the social security system Patient under legal protection Patient suffering from an inflammatory digestive disease Patient on anticoagulant therapy with no possibility of discontinuation or relay Patient with contraindications to colonoscopy/rectosigmoidoscopy Pregnant or breast-feeding patient

Exclusion criteria for control group:

Treatment with anticoagulants Treatment with antiaggregants Subject with a coagulation disorder Subject having finally an abnormal colonoscopy (discovery of any pathology other than one or more benign polyps)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of sulfonic acid and HRP flux in biopsies placed in Ussing chamber | 1 month
Quantifying the expression of junction molecules of the ZO-1 type | 1 month
Number of serotonin-producing cells labelled with anti-5-HT antibody | 1 month
The degree of expression of TPH1 and SERT in RT-qPCR | 1 month
Calculation of the number of neurons and the proportion of different neurochemical phenotypes of neurons in relation to the total number of neurons in the submucosal plexus | 1 month
VIP, ACh and 5-HT concentration in the colonic mucosa | 1 month
Expression levels of key inflammation cytokines (TNFα, IL 1β, IFNɣ...) | 1 month

SECONDARY OUTCOMES:
Correlation between intestinal permeability and type of neurological damage | 1 month
Correlation between intestinal permeability and degree of digestive function impairment | 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nantes service de gastroentérologie, Nantes
  - CHU de Nantes service MPR, Nantes